CLINICAL TRIAL: NCT00941317
Title: A Single-blind Evaluation of Device Performance and Tolerability to Nail Micro-drilling in Subjects With Onychomycosis
Brief Title: Single-blind Evaluation of Device to Nail Micro-drilling in Onychomycosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Michael Graeber, MD, Head of Global Clinical Project Management and US Development, Galderma R&D
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RD.06.CIP.18157
Record Dates: First submitted 2009-07-14; First posted 2009-07-17 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2011-03

CONDITIONS: Onychomycosis
Keywords: onychomycosis; micro-drilling
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pathformer (micro-drilling device) — The micro-drilling device drills the nail with a prespecified diameter drill bit and to a prespecified depth in the nail, using skin impedance (also referred to as equivalent resistivity level) as a feedback mechanism for stopping the drilling intervention at a preset trigger level value.
  Other Names: Pathformer

SUMMARY:
Based on manufacturer testing, no major difference in drilling condition is expected in this study compared to the drilling conditions previously established. However clinical testing is needed to establish optimal drilling conditions to be used for further development in both unaffected and affected parts of the nail. The aim of this study is to determine the optimal drilling condition that could be used in future studies of this device in combination with topical treatment for onychomycosis.

DETAILED DESCRIPTION:
This drug-free, single-blind device study will evaluate the completeness of the holes and the tolerability (pain) of the drilling process by testing several trigger levels. Subjects with distolateral onychomycosis will have a series of holes drilled into the unaffected and affected areas of 1 or 2 big toenail(s). A pain level < 4 using the subject self-assessment Numeric Rating Scale (NRS) is considered as acceptable with regard to the study procedure.

The study will use a two-cohort design in subjects with distolateral onychomycosis.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a male or female 18 years of age or older with clinical diagnosis of distolateral onychomycosis without matrix involvement in at least one big toe with a nail plate at least 2 cm wide. Note: This diagnosis will be based on clinical signs and microscopy; no laboratory culture is required.
* The total disease involvement will be at least 30% and no more than 70% of the total surface of the 1 or 2 big toenail(s) to be drilled in order to allow drilling of up to 5 holes spaced at least 3 mm apart, 5 mm from the lunula, and 2 mm from the lateral edge in each affected and unaffected part of the nail(s).
* The subject is willing and able to comply with the requirements of the CIP and visit schedule. In particular, subjects must agree to remove and not reapply any nail polish or related products to the target toenails for the duration of the study
* The subject understands that this is a drug-free device study for which no therapeutic benefit is expected.
* The subject must agree not to file, clip, or otherwise disturb the target toenail between study visits
* The subject agrees to participate in the study and authorize photographs taken per study requirements, verified by dating and signing an approved written Informed Consent Form (ICF) and Health Insurance Portability and Accountability Act (HIPAA) authorization before any study procedures
* The subject is a female of non-childbearing potential (defined as post-menopausal [absence of menstrual bleeding for 1 year prior to enrollment], hysterectomy or bilateral oophorectomy) or if the subject is a female of childbearing potential and has a negative urine pregnancy test (UPT) at the baseline visit

Exclusion Criteria:

* Affected toenail(s) distal edge of the toenail plate more than 4 mm thick. The distance from the affected distal edge of the toenail plate to the toenail bed will be measured by using a ruler or caliper.
* The subject has other clinically significant nail disease, including clinical signs of nail psoriasis, nail discoloration of nail trauma, or paronychia of the target toenail(s)
* Signs of infection (other than fungal) in one of the feet, including the contralateral foot
* The subject takes daily pain medication, including anti-inflammatory and corticosteroid medications at doses that relieve pain
* The subject takes anti-coagulants (e.g., heparin, warfarin) at therapeutic doses. Prophylactic anti-coagulant therapy (for example inhibitors of platelet aggregation, low dose aspirin, or low molecular weight heparin) is permitted.
* The subject has proximal subungual onychomycosis or only superficial nail plate onychomycosis
* The subject has immunodeficiency, peripheral neuropathy, or peripheral vascular disease, or known types 1 or 2 diabetes.
* The subject has another underlying known disease, a surgical or medical condition that, in the opinion of the Investigator, might interfere with interpretation of the study results
* The subject is currently enrolled in another investigational drug or device study OR participated in such a study in the past 3 months prior to Visit 1 OR in an exclusion period from a previous study
* A female subject is pregnant or plans to conceive a child within 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-07; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Optimize the drilling conditions - to obtain a complete hole and assess tolerability | 1 week

SECONDARY OUTCOMES:
The secondary effectiveness objective is to evaluate the overall performance and reliability of the device | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Alexa B. Kimball, MD, MPH, Principal Investigator — Massachusetts General Hospital, Boston, MA, USA
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States